CLINICAL TRIAL: NCT03863691
Title: Influence of Partial Blockade of Dopaminergic Neurotransmission Using Amisulpride on Stress Responsivity, Motivated Behavior and Emotional Reactivity in Humans.
Brief Title: Influence of Dopaminergic Blockade on Stress Responses, Motivation and Emotional Reactivity in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: III/sja/kno FF96/2018
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Healthy Participants
Keywords: dopamine antagonists; dopamine blockade; psychophysiological stress response; Maastricht acute stress test (MAST); effort based paradigms; positivity offset theory; international affective picture system (IAPS)
MeSH Terms: interventions — Amisulpride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomized, double blind, placebo controlled, between subjects design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- amisulpride group (Active Comparator): 300 mg of the atypical antipsychotic drug amisulpride
  Interventions: Drug: Amisulpride 300 MG
- placebo group (Placebo Comparator): Similar looking capsules for placebo control
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Amisulpride 300 MG — A single dose of 300 mg amisulpride that looks identical to placebo control capsules.
  Arms: amisulpride group
Drug: Placebo oral capsule — A placebo capsule with no inert pharmacological effect. Looks identical to the amisulpride capsules.
  Arms: placebo group

SUMMARY:
The study aims to identify whether partial blockade of human dopamine signaling with antipsychotic drugs affects human stress responses, motivation and emotion. 84 healthy adult participants are planned to complete the study protocol.

Therefore three experiments are planned:

Experiment 1: Influence of amisulpride on human stress responses. Experiment 2: Influence of amisulpride on motivated effort. Experiment 3: Influence of amisulpride on emotion.

DETAILED DESCRIPTION:
The study is a double blind, placebo controlled, randomized trial with two groups. One group will be receiving placebo (PG) and the other group will receive 300 mg amisulpride (VG). All participants are planned to complete all three experiments sequentially after drug/placebo intake.

In experiment 1 we want to test whether a medium single dosage of amisulpride (VG) changes human stress responses compared to the PG. Therefore test subjects take the medication / placebo and wait for peak plasma levels. Afterwards they undergo a standardized stress test (MAST procedure,e.g. Shilton et al., 2017) where they submerge their non-dominant hand in cold water and have to do mental arithmetic tasks. We collect ECG, cortisol and skin conductance data as well as subjective measures of the stress response.

In experiment 2 that is done after completion of experiment 1 the aim is testing whether the VG compared to the PG has an altered motivated effort. Therefore so called effort based paradigms (Reddy et al., 2015) are used. In these paradigms participants are given the option between an easy and effortless way of solving a trial that is reinforced with a small monetary reward or a harder and effortful way of trial solving that is rewarded higher. We measure how often the VG versus the PG will take the easy, low reward option over the hard, high reward option.

In experiment 3 and after the completion of experiment to the aim is it to test whether the mean intensity of visually evoked emotions in the VG is changed compared to the PG. Therefore we use a stimulus set (15 positive images, 15 negative images, 15 neutral images) out of the International Affective Picture System images to evoke emotions and plan to analyze data like in positivity offset research (detailed description in: Strauss et al, 2017).

ELIGIBILITY:
Inclusion Criteria:

* Common European Framework of Reference for Languages level B2 in German language.
* Consent ability for all relevant aspects of the experiment.

Exclusion Criteria:

* Amisulpride allergy.
* Allergy to other components of amisulpride / placebo capsules like lactose.
* Daily intake of other medication including contraceptives.
* Tendency to seizures.
* Diagnosis of cancer especially pheochromocytoma, prolactinoma, or breast cancer.
* Kidney dysfunction: creatinine clearance below 10 ml per minute.
* High risk for stroke or thrombosis.
* Known prolongation of the QT interval,
* Any substantial medical condition that is capable of reducing the volunteers ability to participate at the study.
* Suicidal thoughts or suicide attempts in the past or at present.
* Substantial mental disorders especially schizophrenia, bipolar disorder, drug abuse, or personality disorders.
* Pregnancy or breastfeeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Perceived stress level from baseline to post stress period. | After preparation period. Before (76 min before, 22 min before, 5min before) and after the stress test (directly after, 16 min as well as 30 min after completion).
  Before and after the stress test of experiment 1 we ask every participant for their perceived stress level. These data serve as an indicator of subjective stress responses. We analyze changes in subjective stress level compared to baseline measurements (76 min and 22 min before). Five minutes before the stress test starts we measure subjective anticipatory stress response and directly after the completion we measure post stressor responses and possible residual feelings of stress (16 minutes post completion).
  All measurements reflect a single time series. Stress levels are obtained with visual analogue scales ranging from 0 (no stress) to 100 points (extremely stressed).
Percentage of difficult trials in the balloon effort task. | After the cortisol response of experiment 1 is subsided and directly when experiment is 2 is completely finished. This will be approximately 121 minutes after medication / placebo intake.
  In experiment 2 which is a computer task, participants can choose between an easy task with low monetary reinforcement or a hard task with higher monetary reinforcement. "Easy" means that there is a low amount of physical or cognitive effort per trial and "hard" means that there is a higher amount of physical or cognitive effort per trial. From the tasks that are described in Reddy et al (2015) the balloon effort task (physical effort) and the deck choice task (mental effort) will be used. For both tasks our software automatically obtains the percentage of difficult trials with respect to the total number of trials. Note that only a single composite score is obtained after finishing the balloon effort task.
Percentage of difficult trials in the deck choice task. | After finishing the balloon effort task. This will be approximately 145 minutes after medication / placebo intake.
  In experiment 2 which is a computer task, participants can choose between an easy task with low monetary reinforcement or a hard task with higher monetary reinforcement. "Easy" means that there is a low amount of physical or cognitive effort per trial and "hard" means that there is a higher amount of physical or cognitive effort per trial. From the tasks that are described in Reddy et al (2015) the balloon effort task (physical effort) and the deck choice task (mental effort) will be used. For both tasks our software automatically obtains the percentage of difficult trials with respect to the total number of trials. Note that only a single composite score is obtained after finishing the deck choice effort task.
Mean positive affect ratings in response to International Affective Picture System (IAPS) images. | After experiment 3 is finished. This will be approximately 216 minutes after medication / placebo intake.
  Valence and arousal measures are collected as in Strauss et al. (2017) after presentation of IAPS pictures during experiment 3. Ratings for positive affect, negative affect and arousal ratings are obtained with a 10 point self-assessment manikin scale after the presentation of each individual picture. Note that only a single composite score for positive affect is calculated as the mean value of all evaluations following the individual pictures.
Mean negative affect ratings in response to International Affective Picture System (IAPS) images. | After experiment 3 is finished. This will be approximately 216 minutes after medication / placebo intake.
  Valence and arousal measures are collected as in Strauss et al. (2017) after presentation of IAPS pictures during experiment 3. Ratings for positive affect, negative affect and arousal ratings are obtained with a 10 point self-assessment manikin scale. Note that only a single composite score for negative affect is calculated as the mean value of all evaluations following the individual pictures.

SECONDARY OUTCOMES:
Saliva cortisol levels. | After preparation period. Before (62 min before, 2 min before) and after the stress test (5, 15 and 25 min after completion).
  Before and at three time points after the stress test is completed of experiment 1 we take saliva cortisol samples of each participant. These samples are analysed for cortisol levels and serve as an indicator of Hypothalamic-pituitary-adrenal axis reactivity.
  Cortisol levels are measured in nmol/liter.
Heart rate changes and changes in heart rate variability. | After preparation period. Before (68 min before, 49 min before), during (the whole procedure) and after (directly after completion) the stress test.
  Before, during and after the stress test of experiment 1 we use blood volume pulse measures for obtaining heart rate data and calculate heart rate change scores and heart rate variability scores (HRV). These data serve as an indicator of cardiovascular stress responses.
  Heart rate changes are measured in Δ1/s. Changes in heart rate variability is normalized for heart rate change because higher HR during stress exposure could induce a mathematical bias. Data that will be obtained include the low frequency band and the high frequency / low frequency ratio. A short introduction into the topic can be found in Billmann et al (2015).
Mean arousal ratings in response to International Affective Picture System (IAPS) images. | After experiment 3 is finished. This will be approximately 216 minutes after medication / placebo intake.
  Valence and arousal measures are collected as in Strauss et al. (2017) after presentation of IAPS pictures during experiment 3. Ratings for positive affect, negative affect and arousal ratings are obtained with a 10 point self-assessment manikin scale. Note that only a single composite score for negative affect is calculated as the mean value of all evaluations following the individual pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps-Univeristy of Marburg
Locations (1):
- Clinical Psychology and Psychotherapy, Gutenbergstr. 18, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Billman GE, Huikuri HV, Sacha J, Trimmel K. An introduction to heart rate variability: methodological considerations and clinical applications. Front Physiol. 2015 Feb 25;6:55. doi: 10.3389/fphys.2015.00055. eCollection 2015. No abstract available. PMID 25762937
- [Background] Horan WP, Reddy LF, Barch DM, Buchanan RW, Dunayevich E, Gold JM, Marder SR, Wynn JK, Young JW, Green MF. Effort-Based Decision-Making Paradigms for Clinical Trials in Schizophrenia: Part 2-External Validity and Correlates. Schizophr Bull. 2015 Sep;41(5):1055-65. doi: 10.1093/schbul/sbv090. Epub 2015 Jul 23. PMID 26209546
- [Background] Reddy LF, Horan WP, Barch DM, Buchanan RW, Dunayevich E, Gold JM, Lyons N, Marder SR, Treadway MT, Wynn JK, Young JW, Green MF. Effort-Based Decision-Making Paradigms for Clinical Trials in Schizophrenia: Part 1-Psychometric Characteristics of 5 Paradigms. Schizophr Bull. 2015 Sep;41(5):1045-54. doi: 10.1093/schbul/sbv089. Epub 2015 Jul 3. PMID 26142081
- [Background] Shilton AL, Laycock R, Crewther SG. The Maastricht Acute Stress Test (MAST): Physiological and Subjective Responses in Anticipation, and Post-stress. Front Psychol. 2017 Apr 19;8:567. doi: 10.3389/fpsyg.2017.00567. eCollection 2017. PMID 28469586
- [Background] Strauss GP, Frost KH, Lee BG, Gold JM. THE POSITIVITY OFFSET THEORY OF ANHEDONIA IN SCHIZOPHRENIA. Clin Psychol Sci. 2017 Mar;5(2):226-238. doi: 10.1177/2167702616674989. Epub 2017 Mar 10. PMID 28497008